CLINICAL TRIAL: NCT00747318
Title: A Phase 3, Multicenter, Open-label Continuation Study in Moderate to Severe Asthmatic Subjects Who Completed FlutiForm HFA pMDI Study SKY2028-3-005, Incorporating Amendment 1 and 2
Brief Title: A Phase 3, Multicenter, Open-label Continuation Study in Moderate to Severe Asthmatic Subjects Who Completed FlutiForm HFA pMDI Study SKY2028-3-005
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SkyePharma AG (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Kirsten Kaiser, MD, SkyePharma AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKY2028-3-006
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: Moderate to Severe
MeSH Terms: conditions — Asthma | interventions — fluticasone-formoterol; Fluticasone; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SKP FlutiForm HFA pMDI

INTERVENTIONS:
Drug: SKP FlutiForm HFA pMDI — Each subject will receive SKP FlutiForm HFA pMDI 250/10 microgram twice daily for 60 weeks (two actuations of SKP FlutiForm HFA pMDI 125/5 microgram/actuation) for a total daily dose of 500 microgram fluticasone propionate and 20 microgram formoterol fumarate.
  Other Names: FlutiForm; fluticasone propionate/formoterol fumarate

SUMMARY:
The objective of this study is to assess the long-term safety and efficacy of FlutiForm HFA pMDI 250/10 mcg bid in adolescents and adults with moderate to severe asthma who have completed the study SKY2028-3-005.

ELIGIBILITY:
Inclusion Criteria:

* 1. Documented use of an inhaled corticosteroid for at least 4 weeks prior to the Day 1 (Baseline) visit and at a dose not greater than 500 mcg/day fluticasone propionate inhalation (or equivalent dose for other inhaled corticosteroids). Subjects who enroll in this study SKY2028-3-006 immediately upon completion of study SKY2028-3-005 have automatically satisfied this criterion. Subjects who enroll in this study SKY2028-3-006 after completion of study SKY2028-3-005 within 24 weeks must use inhaled corticosteroid therapy at a dose not greater than 500 mcg/day fluticasone propionate inhalation (or equivalent dose for other inhaled corticosteroids) for at least 4 weeks prior to the Day 1 (Baseline) visit.
* 2. Females of childbearing potential must have a negative urine beta-human chorionic gonadotropin (beta-HCG) pregnancy test at the Day 1 Visit
* 3. Subject is judged to be in good general health as determined by the investigator.
* 4. Demonstrate satisfactory technique in the use of pMDI.

Exclusion Criteria:

* 1. Subjects who prematurely discontinued from the study SKY2028-3-005.
* 2. Life-threatening asthma within the past year.
* 3. History of systemic (oral or injectable) corticosteroid use within the past 12 weeks,
* 4. An upper or lower respiratory infection within 4 weeks prior to the Day 1 (Baseline) visit.
* 5. Significant, non-reversible, pulmonary disease (e.g., chronic obstructive pulmonary disease, cystic fibrosis, bronchiectasis).
* 6. Recent history of smoking, alcohol, substance abuse and/or psychiatric illness,
* 7. Subjects who have taken beta-blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, quinidine type antiarrhythmics, or potent CYP 3A4 inhibitors such as ketoconazole within the past 1 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To assess the long-term safety and efficacy of FlutiForm HFA pMDI 250/10 mcg bid in adolescents and adults with moderate to severe asthma who have completed the study SKY2028-3-005 | week 60

CONTACTS AND LOCATIONS:
Overall Officials: Thao T Doan, MD, Study Director — Abbott Labs PPD R&D
Locations (30):
- United States (10):
  - Investigational Site, Scottsdale, Arizona
  - Investigational Site, Orange County, California
  - Investigational Site, Colorado Springs, Colorado
  - Investigational Site, Valrico, Florida
  - Investigational Site, Elizabeth City, North Carolina
  - Investigational Site, Medford, Oregon
  - Investigational Site, Portland, Oregon
  - Investigational Site, East Providence, Rhode Island
  - Investigational Site, Providence, Rhode Island
  - Investigational Site, West Allis, Wisconsin
- Mexico (5):
  - Investigational Site, Guadalajara, Jalisco
  - Investigational site, Mexico City, Mexico City
  - Investigational Site, Toluca, State of Mexico
  - Investigational Site, Villahermosa, Tabasco Mexico
  - Investigational Site, Zapopan, Zapopan Jalisco
- Investigational site, Lima, Lima Province, Peru
- Romania (6):
  - Investigational site, Constanța, Jud. Constanta
  - Investigational site, Craiova, Jud. Dolj
  - Investigational site, Timișoara, Jud. Timis
  - Investigational site, Bucharest, Sector 1
  - Investigational site, Bucharest, Sector 3
  - Investigational site, Bucharest, Sector 5
- Ukraine (8):
  - Investigational site, Dnipropetrovsk
  - Investigational site, Donetsk
  - Investigational site, Kharkiv
  - Investigational site, Kiev
  - Investigational site, Kyiv
  - Investigational site, Lviv
  - Investigational site, Vinnytsia
  - Investigational site, Zaporizhzhya